CLINICAL TRIAL: NCT04609787
Title: The Effect of Immersive Virtual Reality on Central Sensitization in People With Chronic Pain: A Proof of Concept Pilot
Brief Title: Immersive Virtual Reality and Central Sensitization in People With Chronic Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID prevented acquistion of participants and study funding ended
Sponsor: Tufts University (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Nancy Baker, Associate Professor, Tufts University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000725
Record Dates: First submitted 2020-10-23; First posted 2020-10-30 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain
Keywords: Immersive Virtual Reality
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Pre-IVR MPPTh and MTSP with post IVR levels will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All participants (Experimental): Quantitative sensory testing will be completed and current pain levels obtained. 20-minutes of immersive virtual reality will be completed, and then complete quantitative sensory testing again. We will compare pre-IVR quantitative sensory testing with post IVR levels.
  Interventions: Device: Immersive Virtual Reality

INTERVENTIONS:
Device: Immersive Virtual Reality — Participants are placed in three-dimensional, life-sized computer-generated environments via a computer headset shows potential as a treatment for chronic pain and central sensitization.

SUMMARY:
Patients with chronic low back pain from Dr. Robert Edwards' study at the Brigham & Women's Pain Institute that examines sensory and pain perceptions in patients with chronic pain who use opioids will complete quantitative sensory testing (QST) and current pain levels will be obtained. Subsequently, 20-minutes of Immersive Virtual Reality (IVR) will be completed and then QST testing will be completed again post-IVR.

DETAILED DESCRIPTION:
We will partner with Dr. Robert Edwards at the Brigham & Women's Pain Institute. Dr. Edward's is an expert in testing central sensitization using quantitative sensory testing (QST).12 QST involves cutaneous (skin) psychophysical (semi-subjective) testing to assess sensory and pain perception pathways.13 QST identifies the intensity of stimuli (touch) is needed to feel something (threshold of detection) and how perception of stimuli changes if it is repeated many times (temporal summation).14 In people with central sensitization, even light intensity of stimulation is perceived as pain and similar intensity stimuli becomes more painful with multiple applications. We hypothesize that people with chronic pain will demonstrate clinically important reductions in the threshold of detection and temporal summation after IVR, which will demonstrate that IVR can affect central sensitization.

We will complete two types of QST testing: Mechanical Pressure Pain Thresholds (MPPTh) to test for threshold of detection, and Mechanical Temporal Summation of Pain (MTSP) to test for temporal summation. In MPPTh we will measure the amount of pressure needed at the shoulder and thumb (body sites that routinely do not have pain in people with low back pain) to elicit a pain report from participants. In MTSP we will apply a train of 10 stimuli (light pinprick) at the rate of 1 per second on the middle finger and have participants rate the painfulness of the first, fifth, and tenth stimulus.

During the study, we will recruit 20 patients with chronic low back pain from Dr. Edwards' study examining sensory and pain perceptions in patients with chronic pain who use opioids. We will complete QST testing and obtain current pain levels. We will complete 20-minutes of IVR, and then complete QST testing again. We will compare pre-IVR MPPTh and MTSP with post IVR levels. We anticipate short term, clinically important decreases in QST levels providing initial confirmation that IVR can positively change central sensitization.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-65
2. CLBP lasting for more than 6 months as the primary complaint
3. Typical pain ratings ≥ 4/10 on a visual analogue scale
4. Currently prescribed oral opioid therapy and under consideration for dose reduction by the prescribing clinician.
5. able to speak and understand English

Exclusion Criteria:

1. Evidence of delirium, dementia, psychosis, or other cognitive impairment preventing completion of study procedures
2. current (i.e., active) substance use disorder (SUD).
3. history of myocardial infarction or other serious cardiovascular condition.
4. current peripheral neuropathy.
5. current pregnancy, or intention to become pregnant during the study.
6. current intrathecal pump
7. history of seizures
8. history severe motion sickness

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Quantitative sensory testing (QST): Mechanical Pressure Pain Thresholds (MPPTh) | Completed immediately prior to IVR intervention: Approximately 5 minutes
  Test for threshold of detection: Measure the amount of pressure needed at the shoulder and thumb (body sites that routinely do not have pain in people with low back pain) to elicit a pain report from participants
Quantitative sensory testing (QST): Mechanical Pressure Pain Thresholds (MPPTh) | Completed immediately after IVR intervention: Approximately 5 minutes
  Test for threshold of detection: Measure the amount of pressure needed at the shoulder and thumb (body sites that routinely do not have pain in people with low back pain) to elicit a pain report from participants
Quantitative sensory testing (QST): Mechanical Temporal Summation of Pain (MTSP) | Completed immediately prior to IVR intervention: Approximately 5 minutes
  Test for temporal summation: Apply a train of 10 stimuli (light pinprick) at the rate of 1 per second on the middle finger and have participants rate the painfulness of the first, fifth, and tenth stimulus.
Quantitative sensory testing (QST): Mechanical Temporal Summation of Pain (MTSP) | Completed immediately after IVR intervention: Approximately 5 minutes
  Test for temporal summation: Apply a train of 10 stimuli (light pinprick) at the rate of 1 per second on the middle finger and have participants rate the painfulness of the first, fifth, and tenth stimulus.
PANAS | Completed immediately prior to IVR intervention
  Two scales one for Positive and one for Negative Affect - Score for each scale 10 to 50 with a lower score indicating less of that affect
PANAS | Completed immediately after IVR intervention
  Two scales one for Positive and one for Negative Affect - Score for each scale 10 to 50 with a lower score indicating less of that affect
Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) | Completed immediately prior to IVR intervention
  Scale examining quality of pain with 22 possible pain related symptoms - Score for each scale 0 - 10; 0 as "none", 10 as "worst possible"
Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) | Completed immediately after IVR intervention
  Scale examining quality of pain with 22 possible pain related symptoms - Score for each scale 0 - 10; 0 as "none", 10 as "worst possible"

SECONDARY OUTCOMES:
Simulator Sickness Questionnaire | Completed immediately after IVR experience
  Scale examining symptoms related to user experience in IVR. 16 symptoms. Scale of none, slight, moderate, severe
IGroup Presence Questionnaire | Completed immediately after IVR experience
  User immersion measured with 14 questions related to immersion in IVR experience. Scale of 1-7.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Baker, Principal Investigator — Tufts University
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No